CLINICAL TRIAL: NCT02153203
Title: Using the Prevent-Teach-Reinforce Model to Reduce Problem Behaviors in Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Marc Lanovaz, Assistant Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERFAS-2014-15-058-P
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Autism spectrum disorder; Problem behavior
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autism Spectrum Disorder; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral approach (Experimental): The Prevent-Teach-Reinforce Model will be implemented with families in their home settings.
  Interventions: Behavioral: Prevent-Teach-Reinforce Model
- Educational approach (Active Comparator): Each child's parent will participate in one 2- to 3-hour individual parent training session on the assessment and treatment of problem behavior in children with autism spectrum disorders.
  Interventions: Other: Individual Parent Training Session

INTERVENTIONS:
Behavioral: Prevent-Teach-Reinforce Model — Implementation of the model once to twice per week over a period of 8 weeks
  Arms: Behavioral approach
Other: Individual Parent Training Session — One 2- to 3-hour individual parent training session on the assessment and treatment of problem behavior
  Arms: Educational approach

SUMMARY:
Children with autism spectrum disorders often engage in problem behaviors such as self-injury, destruction, aggression, and stereotypy. Prior research has clearly shown that these problem behaviors may interfere with learning, daily functioning, and social participation. As such, engaging in problem behaviors has a negative impact on the health and quality of life of children with autism spectrum disorders and their families. One promising solution to reduce problem behaviors in this population is the Prevent-Teach-Reinforce (PTR) model, which relies on the evidence-based practices of positive behavior support. Although the use of PTR has been gaining considerably support in schools, the model has never been evaluated as part of a rigorous large-scale study using parents as interventionists. Thus, the purpose of the project is to conduct an assessment of the effectiveness of a home-based version of the PTR model in reducing problem behaviors in children with autism spectrum disorders and in improving families' quality of life. Our hypotheses are that implementing the PTR will (a) produce larger reductions in problem behaviors than participating in an individual parent training session, (b) increase engagement in prosocial behaviors, (c) decrease parental stress, and (c) improve the quality of life of the family. The results of the study will allow an examination of whether PTR is an effective and acceptable model to reduce problem behaviors at home in this population. Given that problem behaviors incur high societal costs when they persist into adolescence and adulthood, the study may potentially lead to large cost reductions in the treatment of difficulties associated with autism spectrum disorders. By reducing engagement in problem behaviors, the implementation of the model may also promote and facilitate the social participation as well as improve the quality of life and health of children with autism spectrum disorders and their families.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorder
* Must exhibit problem behavior

Exclusion Criteria:

* Already receiving services to reduce problem behaviors at home

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parental report of problem behavior at 8 weeks | Prior to the start of the intervention and 8 weeks later
  Problem behavior scale of the Problem Behavior Inventory

SECONDARY OUTCOMES:
Change from baseline in quality of life at 8 weeks | Prior to the start of the intervention and 8 weeks later
  Beach Center Family Quality of Life Scale
Change from baseline in parental report of stress at 20 weeks | Prior to the start of the intervention and 20 weeks later
  Parenting Stress Index Short Form
Change from baseline in parental report of stress at 8 weeks | Prior to the start of the intervention and 8 weeks later
  Parenting Stress Index Short Form
Change from baseline in quality of life at 20 weeks | Prior to the start of the intervention and 20 weeks later
  Beach Center Family Quality of Life Scale
Social validity of the intervention | After 8 weeks of intervention
  Treatment Acceptability Rating Form - Revised
Change from baseline in parental report of problem behavior at 20 weeks | Prior to the start of the intervention and 20 weeks later
  Problem behavior scale of the Problem Behavior Inventory
Change from baseline in parental report of positive social behavior at 20 weeks | Prior to the start of the intervention and 20 weeks later
  Positive social behavior scale of the Nisonger Child Behavior Rating Form
Change from baseline in parental report of positive social behavior at 8 weeks | Prior to the start of the intervention and 8 weeks later
  Positive social behavior scale of the Nisonger Child Behavior Rating Form

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lanovaz, Principal Investigator — Université de Montréal
Locations (3):
- Canada (3):
  - West Montreal Readaptation Centre, Lachine, Quebec
  - CRDITED de Montréal, Montreal, Quebec
  - Gold Centre, Montreal, Quebec